CLINICAL TRIAL: NCT02445352
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Design, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DP-R207 (Rosuvastatin /Ezetimibe Combination) and Rosuvastatin Monotherapy in Patients With Primary Hypercholesterolemia
Brief Title: Efficacy/Safety of DP-R207 Tablet Versus CRESTOR Tablet in Patients With Primary Hypercholesterolemia
Acronym: ROSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP-CTR207-III-02
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Rosuvastatin 5mg & Placebo & Placebo (Active Comparator): Once a day, administration of rosuvastatin 5mg and two types of placebo for 20 weeks
  Interventions: Drug: Rosuvastatin 5mg; Drug: Placebo (for Rosuvastatin 10mg and DP-R207 10/10mg); Drug: Placebo (for Rosuvastatin 20mg and DP-R207 20/10mg)
- DP-R207 5/10mg & Placebo & Placebo (Experimental): Once a day, administration of DP-R207 5/10mg and two types of placebo for 20 weeks
  Interventions: Drug: DP-R207 5/10mg; Drug: Placebo (for Rosuvastatin 10mg and DP-R207 10/10mg); Drug: Placebo (for Rosuvastatin 20mg and DP-R207 20/10mg)
- Rosuvastatin 10mg & Placebo & Placebo (Active Comparator): Once a day, administration of rosuvastatin 10mg and two types of placebo for 20 weeks
  Interventions: Drug: Rosuvastatin 10mg; Drug: Placebo (for Rosuvastatin 5mg and DP-R207 5/10mg); Drug: Placebo (for Rosuvastatin 20mg and DP-R207 20/10mg)
- DP-R207 10/10mg & Placebo & Placebo (Experimental): Once a day, administration of DP-R207 10/10mg and two types of placebo for 20 weeks
  Interventions: Drug: DP-R207 10/10mg; Drug: Placebo (for Rosuvastatin 5mg and DP-R207 5/10mg); Drug: Placebo (for Rosuvastatin 20mg and DP-R207 20/10mg)
- Rosuvastatin 20mg & Placebo & Placebo (Active Comparator): Once a day, administration of rosuvastatin 20mg and two types of placebo for 20 weeks
  Interventions: Drug: Rosuvastatin 20mg; Drug: Placebo (for Rosuvastatin 5mg and DP-R207 5/10mg); Drug: Placebo (for Rosuvastatin 10mg and DP-R207 10/10mg)
- DP-R207 20/10mg & Placebo & Placebo (Experimental): Once a day, administration of DP-R207 20/10mg and two types of placebo for 20 weeks
  Interventions: Drug: DP-R207 20/10mg; Drug: Placebo (for Rosuvastatin 5mg and DP-R207 5/10mg); Drug: Placebo (for Rosuvastatin 10mg and DP-R207 10/10mg)

INTERVENTIONS:
Drug: Rosuvastatin 5mg
  Arms: Rosuvastatin 5mg & Placebo & Placebo
Drug: DP-R207 5/10mg
  Other Names: Rosuvastatin 5mg; Ezetimibe 10mg
  Arms: DP-R207 5/10mg & Placebo & Placebo
Drug: Rosuvastatin 10mg
  Arms: Rosuvastatin 10mg & Placebo & Placebo
Drug: DP-R207 10/10mg
  Other Names: Rosuvastatin 10mg; Ezetimibe 10mg
  Arms: DP-R207 10/10mg & Placebo & Placebo
Drug: Rosuvastatin 20mg
  Arms: Rosuvastatin 20mg & Placebo & Placebo
Drug: DP-R207 20/10mg
  Other Names: Rosuvastatin 20mg; Ezetimibe 10mg
  Arms: DP-R207 20/10mg & Placebo & Placebo
Drug: Placebo (for Rosuvastatin 5mg and DP-R207 5/10mg)
  Arms: DP-R207 10/10mg & Placebo & Placebo; DP-R207 20/10mg & Placebo & Placebo; Rosuvastatin 10mg & Placebo & Placebo; Rosuvastatin 20mg & Placebo & Placebo
Drug: Placebo (for Rosuvastatin 10mg and DP-R207 10/10mg)
  Arms: DP-R207 20/10mg & Placebo & Placebo; DP-R207 5/10mg & Placebo & Placebo; Rosuvastatin 20mg & Placebo & Placebo; Rosuvastatin 5mg & Placebo & Placebo
Drug: Placebo (for Rosuvastatin 20mg and DP-R207 20/10mg)
  Arms: DP-R207 10/10mg & Placebo & Placebo; DP-R207 5/10mg & Placebo & Placebo; Rosuvastatin 10mg & Placebo & Placebo; Rosuvastatin 5mg & Placebo & Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of DP-R207 in patients with primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 19 years
* Signed informed consent form
* At visit 1 and visit 2, LDL-Cholesterol ≤ 250mg/dL and Triglyderide ≤ 350mg/dL

Exclusion Criteria:

* Has a history of hypersensitivity to HMG-CoA reductase inhibitor and component of ezeimibe
* Liver transaminases > 2 x upper limit of normal

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 8 weeks in LDL-Cholesterol | baseline and 8 weeks

SECONDARY OUTCOMES:
Percent change from baseline to 4 weeks in LDL-Cholesterol | baseline and 4 weeks
Percent change from baseline to 4 weeks in lipid related blood test results | baseline and 4 weeks
Percent change from baseline to 8 weeks in lipid related blood test results | baseline and 8 weeks
Percentage of patients reaching treatment goals according to NCEP ATP III Guideline | week 4 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Yangsoo Jang, Ph.D., Study Chair — Severance Hospital
Locations (1):
- Severance Hospital, Seodaemun-gu, Seoul, South Korea